CLINICAL TRIAL: NCT07065045
Title: Psychometric Properties Of Translated Arabic Version Of The Fremantle Shoulder Awareness Questionnaire In Patients With Chronic Shoulder Pain
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, salma khamis mohamed El-gazzar, principal investigator, Cairo University
Other Study IDs: P.T.REC/012/005859
Record Dates: First submitted 2025-06-10; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Chronic Shoulder Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with chronic shoulder pain: Patients with chronic shoulder pain will be aged 18 or more years old . Shoulder pain lasting for more than three months who, after clinical evaluation, will be positive in at least three of the following six clinical tests: (1) Hawkins impingement sign; (2) Neer's impingement sign; (3) painful arc sign; (4) Jobe's test; (5) Whipple's test; (6) shoulder pain elicited by resistance testing during shoulder abduction or external rotation.
  Being conscious and oriented. Able to read and write in Arabic.

SUMMARY:
Test the psychometric properties of translated arabic version of the Fremantle shoulder awareness questionnaire in patients with chronic shoulder pain

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic shoulder pain was aged 18 or more years old .
* Shoulder pain lasting for more than three months which, after clinical evaluation, was positive in at least three of the following six clinical tests: (1) Hawkins impingement sign; (2) Neer's impingement sign; (3) painful arc sign; (4) Jobe's test; (5) Whipple's test; (6) shoulder pain elicited by resistance testing during shoulder abduction or external rotation.
* Being conscious and oriented.
* Able to read and write in Arabic.

Exclusion Criteria:

* History of shoulder surgery or planned shoulder surgery.
* History of fracture, dislocation, or degenerative disease of the shoulder joint.
* Active shoulder range of motion <90 degrees of flexion or abduction or <0 degrees of external rotation.
* Cervical radiculopathy or examination that caused shoulder pain/reduced range of motion after repetitive neck movements.
* Other serious orthopedic problems.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with chronic shoulder pain will be aged 18 or more years old . Shoulder pain lasting for more than three months who, after clinical evaluation, will be positive in at least three of the following six clinical tests: (1) Hawkins impingement sign; (2) Neer's impingement sign; (3) painful arc sign; (4) Jobe's test; (5) Whipple's test; (6) shoulder pain elicited by resistance testing during shoulder abduction or external rotation.
  Being conscious and oriented. Able to read and write in Arabic.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
validity | One week
  questionnaires will be given to chronic painful shoulder patients. Face validity and content validity will be tested by asking physiotherapists who are experienced for > five years if arabic version of the fremantle shoulder awareness questionnaire is easy to use and its contents relevant to the title. construct validity will be tested by applying questionnaires to patients with chronic shoulder pain as gold standard: cross-culturally adapted arabic version of the fremantle shoulder awareness questionnaire(score 0-36, Higher scores indicate greater levels of disturbed bodily self-awareness),Pain Visual Analogue Scale(score 0-100, higher score indicates greater pain intensity), the Quick Disabilities of the Arm, Shoulder and Hand questionnaire(score 0-100 and higher score indicates greater disability),the Shoulder Pain and Disability Index (score 0-10, higher score indicates pain and disability) and the Pain Catastrophizing Scale(score 0-52, higher score indicates high pain perception)
Reliability | one week
  The participants will fill in the Fremantle shoulder awareness questionnaire Arabic version again after 5-7 days without any intervening physical therapy session between those two occasions and at the same time of day to assess the test-retest reliability of the scale. Its overall score ranges from 0-36. Higher scores are associated with greater levels of disturbed bodily self-awareness
feasibility (the time needed to fill out the translated Arabic version of the fremantle shoulder awareness questionnaire.) | one week
  The researcher will calculate the time needed to fill out the translated Arabic version of the fremantle shoulder awareness questionnaire.